CLINICAL TRIAL: NCT02746770
Title: Physiotherapy in Vestibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Physiotherapy Department Coordinator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: vestibularuja
Record Dates: First submitted 2016-02-25; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cawthorne and Cooksey exercises group (Experimental): Intervention: Participants allocated in both control and experimental groups were receiving treatment for their specific vestibular disorders. Patients assigned to the experimental group also performed the Cawthorne and Cooksey exercises for vestibular rehabilitation during a six week of treatment period.
  Interventions: Other: Experimental: Cawthorne and Cooksey exercises group
- control group (No Intervention): intervention: The control group will not perform the active exercise that will be applied to intervention group.

INTERVENTIONS:
Other: Experimental: Cawthorne and Cooksey exercises group — Experimental: intervention group. Patients assigned to the experimental group will perform the Cawthorne and Cooksey exercises for vestibular rehabilitation in addition to their habitual treatment.
  Arms: Cawthorne and Cooksey exercises group

SUMMARY:
Spanish population with unilateral peripheral vestibular disorders.

DETAILED DESCRIPTION:
Participants with peripheral vestibular disorders will be allocated to a Cawthorne and Cooksey exercises protocol or control group. The Cawthorne and Cooksey exercises consist in some head mobilization and positioning tasks which are related with a restoration of vestibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants with with unilateral peripheral vestibular disorders

Exclusion Criteria:

* Bilateral vestibular disorders
* Fluctuating or active unilateral vestibular disease
* Or other medical conditions in the acute phase were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Activities-specific Balance Confidence scale (ABC) | Baseline and after 6 weeks of intervention
  Activities-specific Balance Confidence scale (ABC), to quantify the level of confidence in performing a specific task without losing balance or becoming unsteady. This scale is applied to assess the change due to intervention between the baseline and 6 weeks of treatment. So the data will be collected at baseline and after 6 weeks of treatment.

SECONDARY OUTCOMES:
UCLA Dizziness Questionnaire (UCLA-DQ) | Baseline and after 6 weeks of intervention
  UCLA Dizziness Questionnaire (UCLA-DQ), used to measure the severity and frequency of dizziness and its impact on quality of life. This questionnaire is applied to assess the change due to intervention between the baseline and 6 weeks of treatment. So the data will be collected at baseline and after 6 weeks of treatment.
Dizziness Handicap Inventory (DHI), | Baseline and after 6 weeks of intervention
  Dizziness Handicap Inventory (DHI), to assess the level of disability and handicap.This questionnaire is applied to assess the change due to intervention between the baseline and 6 weeks of treatment. So the data will be collected at baseline and after 6 weeks of treatment.